CLINICAL TRIAL: NCT04974671
Title: Phase II Trial Of Stereotactic Body Radiation Therapy (SBRT) for Oligoprogression on Immune Checkpoint Inhibitors (ICI) in Metastatic Renal Cell Carcinoma
Brief Title: Trial Of Stereotactic Body Radiation Therapy (SBRT) for Oligoprogression on Immune Checkpoint Inhibitors (ICI) in Metastatic Renal Cell Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000027702; No NIH funding (Other: 11.06.23)
Record Dates: First submitted 2021-07-13; First posted 2021-07-23 (Actual); Last update posted 2025-12-04 (Actual); Status verified 2025-12

CONDITIONS: Renal Cell Carcinoma; Metastatic Renal Cell Carcinoma; Oligoprogressive; Progression
MeSH Terms: conditions — Carcinoma, Renal Cell; Disease Progression | interventions — Radiosurgery

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Stereotactic Body Radiation Therapy (Experimental)
  Interventions: Radiation: Stereotactic Body Radiation Therapy

INTERVENTIONS:
Radiation: Stereotactic Body Radiation Therapy — 1-5 fraction Stereotactic Body Radiation Therapy to all sites of progression

SUMMARY:
This Phase II trial will evaluate progression-free survival after Stereotactic Body Radiation Therapy to oligoprogressive (1-5) lesions in metastatic renal cell carcinoma patients on any immune checkpoint inhibitor-containing regimen with last dose of systemic therapy within 3 months prior to trial enrollment.

DETAILED DESCRIPTION:
This Phase II trial will evaluate progression-free survival after Stereotactic Body Radiation Therapy to oligoprogressive (1-5) lesions in metastatic renal cell carcinoma patients on any immune checkpoint inhibitor-containing regimen with last dose of systemic therapy within 3 months prior to trial enrollment. Alternative local therapy (including but not limited to metastectomy or radiofrequency ablation) to one or more of the oligoprogressive lesions is allowed provided at least one of the lesions is receiving Stereotactic Body Radiation Therapy. Stereotactic Body Radiation Therapy will be delivered on nonconsecutive days (if >1 fraction) for a total of 1-5 fractions depending on anatomic site at the treating physicians discretion. Treatment to multiple sites can be delivered sequentially or concurrently, at the treating physicians discretion. Patients will undergo response-assessment imaging (CT chest/abdomen/pelvis with IV contrast and/or PET CT scan and/or MRI plus or minus contrast), and response to treatment will be measured via RECIST. The acute and long-term toxicity will be monitored and graded per CTCAE 5.0 (https://ctep.cancer.gov/). Patients will continue on the same immune checkpoint inhibitor-containing regimen during Stereotactic Body Radiation Therapy planning and delivery, and after completion of Stereotactic Body Radiation Therapy until progression of disease as defined by RECIST criteria. The immune checkpoint inhibitor-containing regimen can be continued beyond RECIST progression of disease if the treating physician feels that a patient will continue to benefit. Each eligible patient will be discussed at a multidisciplinary tumor board in the presence of medical and radiation oncology and will be seen in consultation in a Yale-affiliated radiation oncology department prior to enrollment in the trial.

ELIGIBILITY:
Inclusion Criteria:

In order to be eligible for participation in this trial, the subject must:

1. Be willing and able to provide written informed consent/assent for the trial
2. Be ≥ 18 years of age on day of signing informed consent.
3. Have histologically confirmed renal cell carcinoma with metastatic disease detected on imaging. Biopsy of metastasis is preferred but not required
4. The subject has a performance status of 0, 1, or 2 on the ECOG Performance Scale
5. The life expectancy is > 6 months
6. The most recent systemic therapy must be an ICI-containing regimen, delivered for at least 3 months prior to development of oligoprogressive lesions, with the last dose received within 3 months of trial enrollment.
7. Oligoprogression - defined as documented progression in up to 5 individual lesions with no previous local therapy to those sites using one of the following criteria:

   7.1 RECIST 1.1 7.1.1 At least a 20% increase in the sum of diameters of target lesions (long axis for non-nodal lesions, short axis for nodal lesions), using the previous imaging as a baseline 7.1.2 The sum of all diameters must demonstrate an absolute increase of at least 5 mm 7.1.3 The appearance of at least one new unequivocal lesion 7.2 PERCIST 7.2.1 SUVpeak, normalized to lean body mass (SUL) increase by at least 30% and increase by at least 0.8 SUL of the target lesion 7.2.2 Development of at least one new lesion 7.2.3 Increase in target lesion size by 30% 7.2.4 Unequivocal progression of nontarget lesions 7.3 Progressive enlargement of a known metastasis on 2 consecutive imaging studies at least 2 months apart with a minimum 5 mm increase in size 7.4 Development of a new soft tissue metastatic lesion at least 5 mm in size or any new bone metastasis
8. There is no restriction on the total number of metastases
9. Demonstrate adequate organ function as defined in Table 4, all screening labs should be performed within 28 days of protocol treatment

   Table 4 Adequate Organ Function Laboratory Values

   System Laboratory Value

   Hematological

   Absolute neutrophil count (ANC) ≥ 1,500 /mcL Platelets ≥ 75,000 / mcL Hemoglobin ≥ 9 g/dL

   Renal - IF SBRT will be delivered to a lesion in or abutting the kidney

   Serum creatinine OR ≤1.5 X upper limit of normal (ULN) OR Measured or calculated* creatinine clearance (GFR can also be used in ≥30 mL/min for subject with creatinine place of creatinine or CrCl) levels > 1.5 X institutional ULN

   Hepatic - IF SBRT will be delivered to a lesion in or abutting the liver

   Serum total bilirubin ≤ 1.5 X ULN Direct bilirubin Direct bilirubin ≤ ULN for subjects with total bilirubin levels > 1.5 ULN AST (SGOT) and ALT (SGPT) ≤ 2.5 X ULN OR
   * 5 X ULN for subjects with liver metastases

     * Creatinine clearance should be calculated per institutional standard
10. Able to be treated with SBRT at a Yale radiation oncology facility
11. Female subject of childbearing potential should have a negative urine or serum pregnancy within 72 hours prior to receiving the first dose of SBRT. If the urine test is positive or cannot be confirmed as negative, a serum pregnancy test will be required.
12. Female subjects of childbearing must use an effective form of birth control during this study. Acceptable and highly effective birth control methods include intra-uterine hormone releasing system as well as other methods of birth control including consistent use of an approved oral contraceptive (birth control pill), an implantable contraceptive, an injectable contraceptive, a double-barrier method, or true abstinence. Oral, implantable, or injectable contraceptives are only considered effective if used properly and started at least 30 days prior to the screening visit and continue for 120 days after last dose of study drug. (Reference Section 5.7)
13. Male subjects should agree to use an adequate method of contraception starting with the first dose of study therapy through 6 months after the last dose of study therapy

Exclusion Criteria:

The subject must be excluded from participating in the trial if the subject

1. Has had radiation therapy within 2 weeks of the first protocol treatment.
2. Has brain-only oligoprogression. subjects with brain and systemic oligoprogression can still be considered, however treatment of brain metastases will be per standard of care prior to receiving study SBRT.
3. Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 2 weeks of the first protocol treatment. The use of lowdose steroids for management of chronic conditions is allowed (up to 12mg prednisone orally per day or the equivalent).
4. Has had prior radiation therapy within 2 weeks of the first protocol treatment.
5. Has a known additional malignancy that is progressing or requires active treatment. Exceptions include basal cell carcinoma of the skin, squamous cell carcinoma of the skin, or in situ cervical cancer that has undergone potentially curative therapy.
6. Has an active autoimmune disease requiring systemic treatment within the past 3 months or a documented history of clinically severe autoimmune disease, or a syndrome that requires systemic steroids or immunosuppressive agents. Subjects with vitiligo or resolved childhood asthma/atopy would be an example of an exception to this rule. Subjects that require intermittent use of bronchodilators or local steroid injections would not be excluded from the study. Those with a history of hypothyroidism who are now stable on hormone replacement will not be excluded. Those with Sjorgen's syndrome will not be excluded from the study.
7. Has a history of (non-infectious) pneumonitis that required steroids, current pneumonitis, or underlying lung disease that according to the treating physician makes the patient ineligible.
8. Has an active infection requiring systemic therapy.
9. Is pregnant or breastfeeding, or expecting to conceive or father children within the projected duration of the trial, starting with the screening visit through 120 days after the last dose of trial treatment.
10. Has known active Hepatitis B (e.g., HBsAg reactive) or Hepatitis C (e.g., HCV RNA [qualitative] is detected).
11. Has received a live vaccine within 30 days prior to the first protocol treatment.
12. Has serious medical comorbidities precluding radiotherapy. These include subjects with connective tissue diseases such as lupus or scleroderma, Crohn's disease in subjects where the GI tract will receive radiation
13. Substantial overlap with a previously treated radiation volume. Prior radiotherapy is allowed as long as the composite plan meets dose constraints

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2023-12-22 (Actual); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-04-01 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 6 Months
  The primary objective of this study is to assess progression free survival after SBRT to all sites of progression and continuation of the same systemic regimen in patients with mRCC on ICI-containing systemic regimens with oligoprogression at 1-5 sites. Progression will be defined by RECIST criteria.

SECONDARY OUTCOMES:
Recurrence | Up to two years
  Imaging will be done every three months to determine rate of recurrence.
Rate of Response | Up to two years
  To determine rate of response at non-treated sites. Imaging will be done every three months.
Overall survival | Up to two years
  Overall survival will be assessed up to two years

CONTACTS AND LOCATIONS:
Overall Officials: Kimberly Johung, MD, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No